CLINICAL TRIAL: NCT01817205
Title: A Pilot Study on the Feasibility of Combined Chemoembolization and Adjuvant Systemic Hyperthermia for Palliative Treatment of Unresectable Hepatocellular Carcinoma(HCC)
Brief Title: Combined Chemoembolization and Systemic Hyperthermia for Unresectable Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor case accrual
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other)
Responsible Party: Principal Investigator, Simon Yu, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIR-13-01
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Last update posted 2019-08-30 (Actual); Status verified 2016-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Diathermy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TACE with Hyperthermia treatment (Other): Interventions: TACE to all liver lesions and two sessions of systemic hyperthermia performed at 24 hours and 48 hours respectively after TACE.
  Interventions: Procedure: TACE with Hyperthermia Treatment

INTERVENTIONS:
Procedure: TACE with Hyperthermia Treatment — Transcatheter arterial chemoembolization (TACE) is performed under local anesthesia with right femoral puncture. The feeding lobar hepatic artery is selectively catheterized for drug delivery.
  Systemic hyperthermia is induced with an external energy source using microwave electromagnetic energy, with the patient lying supine on the treatment bed of the hyperthermia equipment, exposing the abdomen to the microwave transmitter.

SUMMARY:
The objective is to evaluate the safety and therapeutic effect of combined hyperthermia and TACE for unresectable HCC

DETAILED DESCRIPTION:
Most patients with Hepatocellular carcinoma (HCC) are diagnosed at an intermediate and advanced stage when the tumors become unresectable. Transcatheter arterial chemoembolization (TACE) has been shown to be effective in prolongation of survival for patients with unresectable HCC and generally adopted as a standard palliative treatment option for patients with intermediate stage HCC. However, the therapeutic effect of TACE in terms of objective tumor response is variable and modest (27%-40%), indicating that there is actually much room for improvement in the treatment. In many cases, patients with intrahepatic HCC uncontrolled after TACE treatment may not be suitable for other treatment options because of their physical condition. For these patients, repeat TACE combined with adjuvant systemic hyperthermia may offer a chance of disease control.

ELIGIBILITY:
Inclusion Criteria:

Patient factor

* Age between 18 and 75
* Child-Pugh A cirrhosis
* Eastern Cooperative Oncology Group(ECOG) performance status Grade 2 or below
* No serious concurrent medical illness
* Prior treatment for HCC including surgery, local ablation, or transarterial treatments allowed
* Imaging evidence of poor intralesional treatment response or disease progression despite transarterial treatment
* Platelet count ≥ 50 10^9/L

Tumor factor

* HCC diagnosed by typical enhancement patterns on cross sectional imaging or histology
* Unresectable and locally advanced disease without extra-hepatic disease
* Hypervascular lesions on CT
* Greatest dimension of the largest tumor ≤15cm

Exclusion Criteria:

Patient factor

* History of significant concurrent medical illness such as ischemic heart disease or heart failure
* Metallic body implants, not including dental fillings
* Serum creatinine level > 130 umol/L
* Presence of biliary obstruction not amenable to drainage
* Child-Pugh B or C cirrhosis
* Unable to give consent

Evidence of impaired liver function

* History of hepatic encephalopathy
* Intractable ascites not controllable by medical therapy
* History of variceal bleeding within last 3 months
* Serum total bilirubin level >25 umol/L for the first 5 patients, serum total bilirubin level >35 umol/L for the second 5 patients
* Serum albumin level < 30g/L
* International normalized ratio(INR) >1.3

Tumor factor

* Presence of extrahepatic metastasis
* Infiltrative lesion

Vascular invasion

* Hepatic artery thrombosis
* Partial or complete thrombosis of the main portal vein
* Tumor invasion of portal branch of contralateral lobe
* Hepatic vein tumor thrombus
* Significant arterioportal shunt
* Significant arteriovenous shunt

Contraindication for hyperthermia

* Known brain metastasis
* Recent stroke or cerebral hemorrhage within last 6 months
* Poorly controlled epilepsy
* Poorly controlled cardiac arrhythmias
* Myocardial infarction within last 6 months
* Unstable angina within last 6 months
* Poorly controlled hypertension
* Poorly controlled diabetes
* History of malignant hyperthermia
* Photodermatosis
* Pregnancy
* Lactation
* Serious infection
* Grade 3 or above adverse event in serological total bilirubin or albumin according to Version 4.0 of National Cancer Institute Common Terminology Criteria for Adverse Events
* Elevation of serum alanine transaminase ≥ 10 times upper limit of normal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
dose limiting toxicity | 30 days from the study treatment

SECONDARY OUTCOMES:
adverse event of treatment | within 6 months of treatment
imaging evidence of objective tumor response | 3 and 6 months after treatment
treatment response by alphafetoprotein | 6 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Simon CH Yu, MD, FRCR, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Imaging and Interventional Radiology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No